CLINICAL TRIAL: NCT03665701
Title: Characterization of the Inhibitory Effects of Fevipiprant (QAW039) on Activation of Eosinophils and ILC2 Cells by Prostaglandin D2 Metabolites
Acronym: 18-03 EONOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18-03 EONOV
Record Dates: First submitted 2018-08-28; First posted 2018-09-11 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Atopic Asthma
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inhibitory effects of Fevipiprant (Experimental): in vitro experiments: The reaction of the innate lymphoid cells by cytokine secretion in response to the stimulation by Prostagalandin D2 metabolites and the measurement of a potential suppressive effect of Fevipiprant will be assessed.
  Interventions: Procedure: Blood Sampling

INTERVENTIONS:
Procedure: Blood Sampling — Blood samples used within in vitro experiments to investigate the activation potency of Prostaglandin D2 metabolites to the DP2 receptor in comparison to Prostaglandin D2.

SUMMARY:
The aim of this study is to draw blood from patients with well-defined atopic asthma that will be subsequently used in invitro experiments to investigate the activation potency of Prostaglandin D2 metabolites to the DP2 receptor in comparison to Prostaglandin D2. The inhibitory activity of a potent DP2 receptor antagonist, Fevipripant, shall be determined.

DETAILED DESCRIPTION:
The inhibitory activity of a potent DP2 receptor antagonist shall be determined. For these experiments eosinophil granulocytes and ILC2 cells will be isolated from the collected blood samples and used in specific assays in respect to their functional reactivity against the DP2 receptor antagonist Fevipiprant after respective stimulation using Prostaglandin D2 metabolites or Prostaglandin D2. Major rationale is to show and determine the EC70 of the effectivity of Fevipiprant against Prostaglandin D2 metabolite triggered activation of eosinophil granulocytes and ILC2 innate lymphoid cells.

ELIGIBILITY:
Inclusion Criteria:

* Women will be considered for inclusion if they are:

Not pregnant, as confirmed by pregnancy test (see flow chart), and not nursing. Of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is pre-menarchial or post-menopausal, with documented proof of hysterectomy or tubal ligation, or meets clinical criteria for menopause and has been amenorrhoeic for more than 1 year prior to the screening visit).

Of childbearing potential and using a highly effective method of contraception during the entire study (vasectomised partner, sexual abstinence - the lifestyle of the female should be such that there is complete abstinence from intercourse from two weeks prior to the first dose of study medication until at least 72 hours after treatment -, implants, injectables, combined oral contraceptives, hormonal IUDs or double-barrier methods, i.e. any double combination of IUD, condom with spermicidal gel, diaphragm, sponge, and cervical cap).

* Body weight ≥ 50 kg and BMI within the range 19-32 kg/m²
* History of allergic asthma since at least 12 months
* A concentration of at least 0,15 x 106/mL eosinophils in peripheral blood

Exclusion Criteria:

* History of an acute infection two weeks prior to the screening visit.
* Intake of oral steroids within 4 weeks prior to screening
* Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, endocrine disease or pulmonary disease (including but not confined to chronic bronchitis, emphysema, tuberculosis, bronchiectasis or cystic fibrosis).
* Participation in another clinical trial 30 days prior to enrollment.
* Donation of more than 100 ml of blood in the preceding 2 months before the screening visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Cytokinesecretion without presence of Fevipiprant | 4 hours after in-vitro exposure of ILC2 cells to prostaglandin D2
  Cytokine release after exposure of ILC2 cells to prostaglandin D2
Cytokinesecretion with presence of Fevipiprant | 4 hours after in-vitro exposure of ILC2 cells to prostaglandin D2
  Cytokine release after exposure of ILC2 cells to prostaglandin D2

CONTACTS AND LOCATIONS:
Locations (1):
- Fraunhofer ITEM im CRC, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No